CLINICAL TRIAL: NCT07284433
Title: A Single-arm, Multicenter, Open-label, Phase I/II Trial of Allo-QuadCAR01-T, an Allogeneic CAR-T-cell Therapy Targeting CD19 and CD20, for the Treatment of Relapsed or Refractory B-cell Malignancies
Brief Title: Study of Allo-QuadCAR01-T, an Allogeneic CAR-T Targeting CD19/CD20, in Patients With Relapsed or Refractory B-Cell Malignancies
Acronym: QUADvance
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AvenCell Therapeutics, Inc. (Industry)
Collaborators: AvenCell Europe GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVC-203-01
Record Dates: First submitted 2025-11-25; First posted 2025-12-16 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma Diffuse Large B-cell; Leukemia and Lymphoma; Leukemia Relapse; Lymphoma Receiving CAR-T Therapy
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Leukemia; Lymphoma | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Intervention Model Description: The trial is structured in three parts: Phase Ia uses a dose-escalation approach to find a safe starting dose of Allo-QuadCAR01-T. Phase Ib expands testing at the selected dose in patients with diffuse large B-cell lymphoma (DLBCL) and possibly other subtypes to confirm safety and early effectiveness. Phase II focuses on a larger group of DLBCL patients to measure how well the treatment works at the recommended dose. All participants receive a single infusion of the therapy after a short course of chemotherapy to prepare their immune system. Patients are closely monitored for 13 weeks, then every three months for two years, with an additional long-term follow-up lasting up to 15 years.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Allo-QuadCAR01-T (Experimental): Phase Ia (Escalation): Participants with relapsed or refractory B-cell malignancies will receive lymphodepleting chemotherapy followed by a single infusion of Allo-QuadCAR01-T.
  Phase Ib (Expansion): After dose escalation, additional participants with relapsed or refractory B-cell lymphoma will receive lymphodepleting chemotherapy followed by a single infusion of Allo-QuadCAR01-T at one or more tolerable dose levels from Phase Ia.
  Phase II: Participants with relapsed or refractory DLBCL will receive lymphodepleting chemotherapy, followed by a single infusion of Allo-QuadCAR01-T at the recommended Phase II dose. The primary endpoint is complete response rate at Week 13, with secondary endpoints including duration of response, progression-free survival, and overall survival.
  Interventions: Other: Cyclophosphamide (Non-IMP, Lymphodepletion); Other: Fludarabine (Non-IMP, Lymphodepletion); Drug: Allo-QuadCAR01-T

INTERVENTIONS:
Other: Cyclophosphamide (Non-IMP, Lymphodepletion) — Intravenous infusion over 3 days (d-5 to d-3)
Other: Fludarabine (Non-IMP, Lymphodepletion) — Intravenous infusion over 3 days (d-5 to d-3)
Drug: Allo-QuadCAR01-T — Single dose IV infusion on Day 1

SUMMARY:
This study is testing Allo-QuadCAR01-T, a new off-the-shelf CAR-T therapy for people with hard-to-treat B-cell cancers. Unlike current CAR-T treatments that use a patient's own cells, this therapy uses donor cells that are ready to use, which can save time and reduce costs. It targets two proteins, CD19 and CD20, to lower the chance of relapse and uses gene editing to make it safer. The trial has three parts: first to find a safe dose, then to confirm it, and finally to test how well it works in patients with diffuse large B-cell lymphoma (DLBCL). Patients will get one infusion after chemotherapy to prepare their body. The main goal is to check safety and see how many patients have a complete response by Week 13. About 160 patients will take part, and researchers will follow them for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older.
* Diagnosed with relapsed or refractory B-cell non-Hodgkin lymphoma (B-NHL) or chronic lymphocytic leukemia (CLL).
* Must have received at least 2 prior lines of therapy.
* ECOG performance status 0-1 (able to carry out daily activities).
* Adequate organ function (heart, liver, kidneys).
* HLA B/C match with donor cells.
* No active uncontrolled infections.

Exclusion Criteria:

* Active CNS involvement (including PCNSL) in dose escalation cohorts; may be allowed in later cohorts with Sponsor approval.
* Prior CAR-T within 3 months of screening, or ≥Grade 3 ICAHT from prior CAR-T.
* Autologous stem cell transplant within 3 months.
* Prior allogeneic stem cell transplant or solid organ transplant.
* Prior therapy with dual CD19/CD20 CAR-T.
* Severe hypersensitivity to trial agents or similar compounds.
* History of GvHD or post-transplant lymphoproliferative disorder.
* Presence of La/SS-B autoantibodies or related autoimmune diseases.
* Other malignancy that may interfere with trial, except:

  * Curatively treated basal/squamous skin cancer or cervical carcinoma in situ
  * Low-grade, early-stage prostate cancer (Gleason ≤6, Stage 1-2) with no therapy needed
  * Adjuvant endocrine therapy for non-metastatic breast cancer (≥2 years)
  * Any other curatively treated malignancy in remission ≥2 years
* Active viral infection within 1 week of screening, or serious bacterial/fungal infection.
* Hemorrhagic cystitis.
* Active neuro-autoimmune disease (e.g., MS, Guillain-Barré, ALS).
* Active or residual HBV, HCV, or syphilis.
* Active HIV. History of HIV may be eligible with Sponsor approval if:
* Neurological disorders within 6 months (e.g., stroke, dementia, Parkinson's, cerebellar disease, CNS autoimmune disease).
* Significant cardiac disease within 6 months (e.g., MI, stent, unstable angina).
* Primary immunodeficiency or autoimmune disease requiring systemic treatment within 1 year (unless stable and Sponsor-approved).
* Unresolved ≥Grade 2 non-hematologic toxicity from prior therapy (except neuropathy up to Grade 2).
* Systemic immunosuppression within 28 days.
* Last systemic lymphoma/CLL therapy (standard or investigational) within 28 days or 5 half-lives.
* Major surgery within 14 days.
* Local radiation within 28 days.
* Live vaccination within 28 days.
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2029-04-27 (Estimated); Study Completion 2029-11-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs defined as DLTs | At the end of cycle 1 (in total 28 days, given no treatment interruptions)
  Incidence and intensity of adverse events (AEs) graded according to Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0, except for cytokine release syndrome (CRS), immune effector cell associated neurotoxicity syndrome (ICANS), tumor lysis syndrome, and graft versus host disease (GvHD), which will be graded according to widely accepted specialized criteria
To determine the maximum tolerated dose (MTD) | At the End of Cycle 1 (in total 28 days, given no treatment interruptions)
  MTD
To determine the incidence of dose-limiting toxicities (DLT) | At the end of cycle 1 (in total 28 days, given no treatment interruptions)
  Incidence of DLTs
Phase 2: Complete response rate (CRR) | Up to week 13
  Complete remission rate is defined as the proportion of participants with complete remission, per international working group (IWG) Lugano classification, as assessed by the investigator.

SECONDARY OUTCOMES:
Pharmacokinetics of Allo-QuadCAR01-T in PB in patients after infusion of Allo-QuadCAR01-T | Up to 24 months
  Detection of VCN in blood samples
To investigate the impact of Allo-QuadCAR01-T on MRD | Up to 24 months
  MRD levels in responding CLL patients
To evaluate immunogenicity against Allo-QuadCAR01-T | Up to 24 months
  Incidence of ADA1 formation against anti-CD19/CD20 ECD and ADA2 formation against the RevCAR ECD of Allo-QuadCAR01-T
To evaluate host immune cell depletion and reconstitution resulting from LD | Up to 24 months
  Enumeration of host PB B-cell, T cell, and NK cell numbers
Overall Response Rate (ORR) | Up to 24 months
  ORR is defined as the proportion of participants with best objective response of either a CR or a partial response (PR) during the trial prior to any new anti-lymphoma, anti-CLL therapy or local radiotherapy for lymphoma , per the Lugano Classification, as determined by the investigator.
Progression-Free Survival (PFS) | Up to 24 months
  PFS is defined as the time from Allo-QuadCAR01-T infusion to disease progression per the Lugano Classification, as determined by investigator review or death from any cause.
Duration of Response (DOR) | Up to 24 months
  DOR is defined as the time from first objective response to disease progression or death from any cause among participants who have achieved CR or PR per the Lugano Classification, as determined by the investigator.
Overall Survival (OS) | Up to 24 months
  OS is defined as the time from Allo-QuadCAR01-T infusion to death from any cause.
Time to Next Treatment (TTNT) | Up to 24 months
  TTNT is defined as time from Allo-QuadCAR01-T infusion to the start of subsequent new anti-lymphoma, anti-CLL therapy or local radiotherapy for lymphoma.

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (6):
  - Universitatsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen, Erlangen, Bavaria
  - Klinikum der Universität München, Munich, Bavaria
  - Universitätsklinikum Marburg, Marburg, Hesse
  - Universitätsklinikum Dresden, Dresden, Saxony
  - Charité Universitätsmedizin Berlin, Berlin